CLINICAL TRIAL: NCT03077165
Title: A 10-week Randomized, Double-blind, Placebo-controlled, Prospective, International, Multicentre, Phase IIa Study of S42909 on Leg Ulcer Healing.
Brief Title: Dose-response Relationship Study of S42909 on Leg Ulcer Healing
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ilkos Therapeutic Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL2-42909-016
Record Dates: First submitted 2017-03-01; First posted 2017-03-10 (Actual); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group A (Experimental): S42909 dose 100 mg p.o., 50 mg bid
  Interventions: Drug: S42909 100 mg
- Group B (Experimental): S42909 dose 200 mg p.o., 100 mg bid
  Interventions: Drug: S42909 200 mg
- Group C (Experimental): S42909 dose 400 mg p.o., 200 mg bid
  Interventions: Drug: S42909 400 mg
- Group D (Experimental): S42909 dose 800 mg p.o., 400 mg bid
  Interventions: Drug: S42909 800 mg
- Group E (Experimental): S42909 dose 1200 mg p.o., 600 mg bid
  Interventions: Drug: S42909 1200 mg
- Group F (Placebo Comparator): Placebo p.o. bid
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: S42909 100 mg — 50 mg Film-coated tablets per os administration, twice a day taken at the end of the morning and at evening meals.
  Arms: Group A
Drug: S42909 200 mg — 50 mg Film-coated tablets per os administration, twice a day taken at the end of the morning and at evening meals.
  Arms: Group B
Drug: S42909 400 mg — 200 mg Film-coated tablets per os administration, twice a day taken at the end of the morning and at evening meals.
  Arms: Group C
Drug: S42909 800 mg — 200 mg Film-coated tablets per os administration,twice a day taken at the end of the morning and at evening meals.
  Arms: Group D
Drug: S42909 1200 mg — 200 mg Film-coated tablets per os administration, twice a day taken at the end of the morning and at evening meals.
  Arms: Group E
Drug: Placebo Oral Tablet — Matching placebo tablets, per os administration, twice a day taken at the end of the morning and at evening meals.
  Arms: Group F

SUMMARY:
Dose-response relationship study of S42909 on leg ulcer healing after oral repeated administration in patients with active venous leg ulcer.

DETAILED DESCRIPTION:
S42909 is an inhibitor of β-Nicotinamide Adenine Dinucleotide Phosphate (NADPH) oxidase which also inhibits vascular leukocyte adhesion to endothelial cells, Matrix Metalloproteinase-2 (MMP-2) and Plasminogen Activator Inhibitor-1 (PAI-1) activity. It is proposed for development in the treatment of venous and mixed leg ulcers.

This proof of concept study is a randomized, double-blind, placebo-controlled, multicenter, Phase IIa trial to evaluate the dose response of S42909 for the treatment of venous leg ulcers.

Patients suffering from chronic venous disease and having at least one active venous leg ulcer will be selected at the selection visit (ASSE). One Reference Ulcer (RU) defined as the largest ulcer in size that is fitting the area selection criteria will be established. At ASSE, a first picture will be taken before cleansing and debridement and a second picture will be taken after cleansing and debridement. The investigator will check that the selection RU area is compliant with the selection criteria. Patients will start the selection period and will be switched from their current pharmacological and/or local treatment (if any) for venous leg ulcer to local wound care with sterile saline solution or sterile water, "non-active" dressings and standardized compression (same strength and type of compression). They will be administrated the placebo selection treatment for a period of fourteen days.

Three (or four) working days before the inclusion visit, the participants will come to the site for a RU picture in order to get the RU area central measurement for inclusion visit (W000).

At W000, the investigator will check that the inclusion RU area is compliant with the inclusion criteria. The investigator will also check that the participant is compliant with the selection treatment and stockings wearing.

All participants found to be eligible for inclusion will be randomized to one of the following six groups - S42909: 100, 200, 400, 800 or 1200 mg per day- or placebo.

The participants will enter a 6 weeks ambulatory Investigational Medicinal Product (IMP) treatment period on top of standard of care (standardized compression and local wound care with sterile saline solution or sterile water and "non-active" dressing) followed by a 2 weeks follow-up period of standard of care only. During this period the participants will return to the investigator's site for intermediate visits after one week (W001), two weeks (W002), three weeks (W003), four weeks (W004), six weeks (W006) and eight weeks (W008). Participants will continue receiving standardized compression therapy and local wound care (sterile saline solution or sterile water and "non-active" dressing) until the end of the study (W008).

ELIGIBILITY:
Inclusion Criteria:

* Caucasian (defined for this study as having 2 Caucasian parents), men or women
* Age ≥ 18 years old
* 18.5 kg/m2 ≤ BMI ≤ 45.0 kg/m2 (= Weight (kg) / height² (m²))
* Patients with chronic venous disease documented by imaging to detect a venous disorder in one or both the sub- and extra-fascial venous systems. The examination performed within 6 months before selection can be used.
* Patients with at least one active venous leg ulcer localised in the gaiter area (CEAP C6) diagnosed or reoccurred for more than 6 weeks and less than 2 years at selection and 3 cm away from other ulcers. Patients with bilateral ulcerations or multiple ulcerations on one or both legs are eligible for selection.
* Size of Reference Ulcer (defined as the largest ulcer in size that is fitting the area selection criteria) should be ≥ 5 cm2 and ≤ 100 cm2 at the selection visit and ≥ 4.5 cm2 and ≤ 100 cm2 at the inclusion visit (measured by transparent sheet and confirmed with the digital 3D imaging device).
* Ankle Brachial Pressure Index (ABPI) ≥ 0.8 and ≤ 1.3 measured by Doppler ultrasound.

Exclusion Criteria:

* Unlikely or unwilling to be compliant to standardized compression recommendation, study medication and visits, previous records of poor compliance to compression stockings.
* Inadequately controlled type 1 and type 2 diabetes with an HbA1c > 8%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2020-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eberhard Rabe, Professor, Principal Investigator — Department of Dermatology University of Bonn
Locations (80):
- United States (14):
  - ILD Research Center, Carlsbad, California
  - Center for Clinical Research Inc., Carmichael, California
  - Center for Clinical Research Inc., Castro Valley, California
  - Limb Preservation Platform, Inc., Fresno, California
  - Foot and Ankle Clinic, Los Angeles, California
  - Stanford Hospitals and Clinics, Redwood City, California
  - Center for Clinical Research Inc., San Francisco, California
  - University of Miami Hospital Wound Center, Miami, Florida
  - St. Luke's Intermountain Research Center, Boise, Idaho
  - Podiatry 1st, Belleville, Illinois
  - Advanced Foot & Ankle Center, Las Vegas, Nevada
  - The Snyder Institute for Vascular Health and Research, Kittanning, Pennsylvania
  - D&P Medical Group, LLC, Pittsburgh, Pennsylvania
  - Serena Group Research Foundation, Pittsburgh, Pennsylvania
- Argentina (4):
  - Centro Dr Bottini de flebologia y estetica, Ciudad Autonoma de Buenos Aire
  - Hospital Italiano de La Plata, La Plata
  - DIM Clinica Privada, Ramos Mejía
  - Sanatorio Mapaci, Rosario
- Austria (3):
  - Medizinische Universitaet Innsbruck Universitaetsklinik für Gefässchirurgie, Innsbruck
  - VENEX Zentrum fuer minimal invasive Venentherapie, Vienna
  - Medizinische Universitaet Wien AKH- Dermatologie, Vienna
- Brazil (6):
  - Faculdade de Medicina de Botucatu, Botucatu
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - Faculdade de Medicina do ABC Cepes, Santo André
  - Centro Multidisciplinar de Estudos Clinicos CEMEC, São Bernardo do Campo
  - Hospital Sao Paulo, São Paulo
  - Hospital Sao Vicente de Paulo, Teixeira Soares
- Canada (7):
  - Alberta Health Services, Calgary, Alberta
  - Parkwood Institute, London, Ontario
  - Toronto Regional Dermatology & Wound Healing Clinic, Mississauga, Ontario
  - Ottawa Hospital Civic Campus, Ottawa, Ontario
  - Centrepoint Medical Center, Ottawa, Ontario
  - York Dermatology Center, Richmond Hill, Ontario
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
- Czechia (5):
  - I. Dermatovenerologicka Klinika, Brno
  - MATMED s.r.o., Hodonín
  - Nemocnice Jihlava Chirurgie A, Jihlava
  - Nemocnice Trebic Kozni oddeleni p.o., Třebíč
  - Angiocor s.r.o., Zlín
- Hungary (10):
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Peterfy Sandor Utcai Korhaz, Budapest
  - Egyesitett Szent Istvan es Szent, Budapest
  - Bajcsy-Zsilinsky Korhaz, Budapest
  - Magyar Honvedseg Egeszsegugyi, Budapest
  - Debreceni Egyetem Orvos es Egeszsegtudomanyi Centrum, Debrecen
  - Bacs-Kiskun Megyei Korhaz, Kecskemét
  - Josa Andras Oktatokorhaz, Nyíregyháza
  - Pesi Tudomanyegyetem Klnikai Kozpont, Pécs
  - Szegedi Tudomanyegyetem Borgyogyaszati es Allergologiai Klinica, Szeged
- Italy (8):
  - Azienda Ospedaliera San Giuseppe Moscati Medicina interna, Avellino
  - Ospedale San Bassiano - Azienda ULSS n. 7 Pedemontana - Ambulatorio di Vulnologia, Bassano del Grappa
  - Ospedale San Giacomo Apostolo Castelfranco Veneto - U.O. Angiologia, Castelfranco Veneto
  - Policlinico Vittorio Emanuele - Presidio Ospedaliero Vittorio Emanuele, Catania
  - Azienda Ospedaliero Universitaria di Padova U.O. Angiologia - Medicina Vascolare, Padua
  - Istituto Neurologico Mediterraneo NEUROMED U.O.C. Chirurgia Vascolare ed Endovascolare, Pozzilli
  - Ospedale Basso Ionio ASPCZ U.O.C. Chirurgia Generale, P.O. di Soverato, Soverato Marina
  - Ospedale Belcolle - U.O Angiologia, Viterbo
- Poland (5):
  - ClinicMed Daniluk, Bialystok
  - Szpital Uniwersytecki nr 1 im. Antoniego Jurasza, Bydgoszcz
  - Medical Academy of Lublin, Lublin
  - SP Szpital Kliniczny Nr1, Poznan
  - Klinika Flebologii, Warsaw
- Slovakia (10):
  - ALIAN, s.r.o., Poliklinika ČK plus, Bardejov
  - BeneDerma, Bratislava
  - Derm-Therapy, Bratislava
  - M.M.-Angio spol. s r.o., Angiologicka ambulancia, Dunajská Streda
  - ANGIOCARE, s.r.o., Košice
  - ALIAN, s.r.o., Angiologická ambulancia, Poprad
  - Dermatovenerologicke oddelenie SANARE, spol. s r.o., Svidník
  - Nemocnica arm. generala L. Svobodu Svidnik, Svidník
  - MEDENA s.r.o., Angiologicka ambulancia, Trnava
  - MEDIVASA, s.r.o., Žilina
- Spain (8):
  - Fundacion Hospital de Aviles, Avilés
  - Hospital Vall d'Hebron, Barcelona
  - Consorci Sanitari de Terrassa - Hospital de Terrassa, Barcelona
  - Hospital Universitario de Getafe, Getafe
  - Hospital de la Cruz Roja de Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Complejo Asistencial Universitario, Salamanca
  - Hospital de Manises, Valencia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A | Group B | Group C | Group D | Group E | Group F
Started | 21 | 22 | 20 | 19 | 19 | 20
Completed | 20 | 22 | 20 | 19 | 16 | 20
Not Completed | 1 | 0 | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A: S42909 dose 100 mg p.o., 50 mg bid
  S42909 100 mg: 50 mg Film-coated tablets taken orally, twice a day taken at the end of the morning and at evening meals.
- Group B: S42909 dose 200 mg p.o., 100 mg bid
  S42909 200 mg: 50 mg Film-coated tablets taken orally, twice a day taken at the end of the morning and at evening meals.
- Group C: S42909 dose 400 mg p.o., 200 mg bid
  S42909 400 mg: 200 mg Film-coated tablets taken orally, twice a day taken at the end of the morning and at evening meals.
- Group D: S42909 dose 800 mg p.o., 400 mg bid
  S42909 800 mg: 200 mg Film-coated tablets taken orally,twice a day taken at the end of the morning and at evening meals.
- Group E: S42909 dose 1200 mg p.o., 600 mg bid
  S42909 1200 mg: 200 mg Film-coated tablets taken orally, twice a day taken at the end of the morning and at evening meals.
- Group F: Placebo p.o. bid
  Placebo Oral Tablet: Matching placebo tablets taken orally, twice a day taken at the end of the morning and at evening meals.
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Group D | Group E | Group F | Total
Number analyzed (Participants) | 21 | 22 | 20 | 19 | 19 | 20 | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 12 | 12 | 4 | 9 | 11 | 57
  >=65 years | 12 | 10 | 8 | 15 | 10 | 9 | 64
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 10 | 13 | 14 | 10 | 66
  Male | 11 | 13 | 10 | 6 | 5 | 10 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 21 | 22 | 20 | 19 | 19 | 20 | 121
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Argentina | 0 | 4 | 1 | 2 | 2 | 2 | 11
  Hungary | 2 | 2 | 1 | 0 | 2 | 1 | 8
  United States | 1 | 1 | 2 | 1 | 2 | 1 | 8
  Czechia | 4 | 4 | 4 | 5 | 4 | 5 | 26
  Spain | 2 | 2 | 1 | 1 | 3 | 2 | 11
  Canada | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Austria | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Brazil | 3 | 3 | 2 | 2 | 1 | 2 | 13
  Poland | 1 | 0 | 0 | 1 | 0 | 0 | 2
  Italy | 2 | 2 | 2 | 3 | 2 | 2 | 13
  Slovakia | 5 | 4 | 6 | 4 | 3 | 4 | 26

OUTCOME MEASURES:

1. Primary Outcome: Relative Reduction of Reference Ulcer Area After 4 Weeks of Treatment on Top of Standard of Care Compared With Baseline Reference Ulcer Area (W000) Assessed During Study Visits
Description: Change of reference Ulcer area measurement in cm^2 from Baseline to Week 4.
Time Frame: Baseline and Week 4
Measure: Geometric Mean (Standard Deviation); unit: cm2
Arm/Group | Group A | Group B | Group C | Group D | Group E | Group F
Number analyzed (Participants) | 20 | 22 | 20 | 19 | 19 | 20
cm2 | -52.85 (37.79) | -46.42 (33.30) | -31.07 (38.73) | -43.33 (28.37) | -41.10 (33.99) | -41.23 (43.71)

2. Secondary Outcome: Adverse Events
Description: Occurring during the double-blind period of the study
Time Frame: Up to 8 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Assessment of Laboratory Parameters
Description: Biochemistry, Haematology and Fasting Lipids
Time Frame: Up to 8 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each participants from the Selection visit (day -14) through end of study visit (Week 8) which is approximately during 10 weeks.
Arm/Group | Group A | Group B | Group C | Group D | Group E | Group F
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22 | 0/20 | 0/19 | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 2/21 | 0/22 | 1/20 | 1/19 | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 4/21 | 6/22 | 8/20 | 6/19 | 8/19 | 6/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=21) | Group B (N=22) | Group C (N=20) | Group D (N=19) | Group E (N=19) | Group F (N=20)
Hypertension (Vascular disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0
Cardiac Failure (Cardiac disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0
Pneumonia (Infections and infestations) | 1 (1) | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=21) | Group B (N=22) | Group C (N=20) | Group D (N=19) | Group E (N=19) | Group F (N=20)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incorrect product administration duration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
C-reactine protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltrnasferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increased bronchial secretions (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (4) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pseudopolyposis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritis generalized (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 2 (4) | 1 (2) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyploglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-03-05): https://cdn.clinicaltrials.gov/large-docs/65/NCT03077165/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT03077165/SAP_001.pdf